CLINICAL TRIAL: NCT02822625
Title: Efficacity of a Standardized Hypnotic Message on Pain Experienced During the Application of a Qutenza (Capsaicin) 8% Patch in Patients With Peripheral Neuropathic Pain
Brief Title: Efficacity of a Standardized Hypnotic Message During the Application of a Qutenza (Capsaicin) 8% Patch
Acronym: ENHYZA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A00234-47
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pain
Keywords: Capsaicin; QUTENZA®; Hypnosis; Peripheral Neuropathic
MeSH Terms: conditions — Pain; Neuritis | interventions — Capsaicin; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- arm 1 (Experimental): Patients, followed in the institut and for whom a new application of QUTENZA® is required, will receive standard care.
  Interventions: Drug: QUTENZA®
- arm 2 (Active Comparator): Patients, followed in the institut and for whom a new application of QUTENZA® is required.
  Patients will receive QUTENZA® according to standard procedure with a standardized hypnotic message
  Interventions: Drug: QUTENZA®; Other: hypnotic message
- arm 3 (Placebo Comparator): Patients, followed in the institut and for whom a new application of QUTENZA® is required.
  Patients will receive QUTENZA® according to standard procedure with a music therapy
  Interventions: Drug: QUTENZA®; Other: music therapy

INTERVENTIONS:
Drug: QUTENZA®
Other: hypnotic message
  Arms: arm 2
Other: music therapy
  Arms: arm 3

SUMMARY:
QUTENZA® is a skin patch with a high concentration of capsaicin (8%) which is the component responsible for spicy peppers. QUTENZA® is indicated for the treatment of peripheral neuropathic pain in non-diabetic adults either alone or in combination with other analgesics. Acute pain experienced during and after the procedure can be relieved by local cooling methods and oral analgesics but the pain remains intense. The hypothesis is that hypnosis via a standardized hypnotic message would increase the local tolerance of the treatment when applying the patch QUTENZA®. To date, there are no studies that can confirm or refute this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have already received at least a QUTENZA® patch
* Treatment for patient in failure to conventional treatments for neuropathic pain other than diabetics
* Age >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <3
* Patient must be affiliated to a social security system
* Ability to provide written informed consent
* Patient's legal capacity to consent to study participation and to understand and comply with the requirements of the study

Exclusion Criteria:

* Patient with psychotic disorders
* Patient with hearing disorders
* Patient not understanding the French language
* Age < 18 years
* Patient requiring analgesic premedication before applying the patch QUTENZA®
* Patient with a history of hypersensitivity to capsaicin or any of the excipients of the patch
* Patient deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Compare pain induced by patch QUTENZA® | 1 day
  Pain will be evaluated by a numerical scale before, just after, and after installation of the patch

SECONDARY OUTCOMES:
Compare anxiety induced by patch QUTENZA® | 1 day
  Anxiety will be evaluated by a numerical scale before, just after, and after installation of the patch
Compare the real time of application of the patch | 1 day
Determine the number of patients who listened the message in totality. | 1 day
Compare the percentage of patients with a sensation of time distortion | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: CRETINEAU Nathalie, Md, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Etienne R, Laurent M, Henry A, Bioy A, Salleron J, Schohn CH, Cretineau N. Interest of a standardized hypnotic message for the reduction of pain and anxiety in cancer patients treated by capsaicin patch for neuropathic pain: a randomized controlled trial. BMC Complement Med Ther. 2021 May 27;21(1):154. doi: 10.1186/s12906-021-03329-8. PMID 34044838